CLINICAL TRIAL: NCT06337578
Title: Avanzamenti in Materia di Screening Cognitivo Telefonico
Brief Title: Advances in Telephone-based Cognitive Screening Procedures
Acronym: TBCS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C308
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Alzheimer's Disease; Lewy Body Dementia; Frontotemporal Degeneration; Cerebrovascular Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Alzheimer Disease; Lewy Body Disease; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with amyotrophic lateral sclerosis (ALS): Individuals having been received a clinical diagnosis of amyotrophic lateral sclerosis according to current diagnostic criteria
  Interventions: Behavioral: Telephone-based neuropsychological assessment - ALS
- Patients with Alzheimer's disease (AD): Individuals having been received a neurochemical and/or aclinical diagnosis of Alzheimer's according to current diagnostic criteria
  Interventions: Behavioral: Telephone-based neuropsychological assessment - AD, LBD, FTD and CVD
- Patients with Lewy body dementia (LBD): Individuals having been received a clinical diagnosis of Lewy body dementia according to current diagnostic criteria
  Interventions: Behavioral: Telephone-based neuropsychological assessment - AD, LBD, FTD and CVD
- Patients with frontotemporal dementia (FTD): Individuals having been received a clinical diagnosis of frontotemporal dementia (i.e., behavioural variant-frontotemporal dementia; semantic dementia; progressive non-fluent aphasia) according to current diagnostic criteria
  Interventions: Behavioral: Telephone-based neuropsychological assessment - AD, LBD, FTD and CVD
- Patients with chronic cerebrovascular disorders (CVD): Individuals with mild cognitive impairment/dementia and neuroradiological evidence of chronic cerebrovascular diseases
  Interventions: Behavioral: Telephone-based neuropsychological assessment - AD, LBD, FTD and CVD
- Normotypical individuals (NI): Individuals without brain disorders
  Interventions: Behavioral: Telephone-based and in-person cognitive screening - NIs

INTERVENTIONS:
Behavioral: Telephone-based neuropsychological assessment - ALS — ALS patients will be administered the following TBCS tests:
  * ALS Cognitive Behavioral Screen-Phone Version;
  * Telephone-based Frontal Assessment Battery;
  * Telephone Language Screener;
  * Telephone-based Verbal Fluency Battery;
  This group will also undergo a telephone-based, caregiver-reported behavioral and functional assessment via the following scales:
  * Activities of Daily Living;
  * Instrumental Activities of Daily Living;
  * Amsterdam IADL Questionnaire - Short Version;
  * Caregiver Behavioral Questionnaire;
  * ECAS-Carer Interview.
  Groups: Patients with amyotrophic lateral sclerosis (ALS)
Behavioral: Telephone-based neuropsychological assessment - AD, LBD, FTD and CVD — AD, DLB, FTD and CVD patients will be administered the following TBCS tests:
  * Telephone Interview for Cognitive Status;
  * Telephone-based Frontal Assessment Battery;
  * Telephone Language Screener;
  * Telephone-based Verbal Fluency Battery;
  These groups will also undergo a telephone-based, caregiver-reported behavioral and functional assessment via the following scales:
  * Activities of Daily Living;
  * Instrumental Activities of Daily Living;
  * Amsterdam IADL Questionnaire - Short Version;
  * Neuropsychiatric Inventory;
  * Frontal Behavioural Inventory.
  Groups: Patients with Alzheimer's disease (AD); Patients with Lewy body dementia (LBD); Patients with chronic cerebrovascular disorders (CVD); Patients with frontotemporal dementia (FTD)
Behavioral: Telephone-based and in-person cognitive screening - NIs — NIs will undergo the Telephone Interview for Cognitive Status over the telephone and will be additionally administered, in person, the following cognitive screeners:
  * Mini-Mental State Examination
  * Montreal Cognitive Assessment
  * In-Person Telephone Interview for Cognitive Status in person.
  Groups: Normotypical individuals (NI)

SUMMARY:
1. Background

   Cognitive screening procedures via performance-based tests represent an essential, albeit preliminary, element within the diagnostic and interventional process as addressed to patients with chronic neurological disorders. Furthermore, in these populations, cognitive screening measures are often employed as outcomes in epidemiological settings, as well as endpoints in clinical trials. Therefore, cognitive screeners need to possess robust clinimetric and clinical usability properties - the investigation of which must be country-specific (i.e., specific to each language and culture).

   The need for such clinimetric and feasibility studies is even more true if referred to telephone-based cognitive screening (TBCS) procedures - which, until recently, have been mostly neglected in Italy, despite having the potential to bring clear benefits to clinical practice and research. In fact, TBCS techniques allow, through the use of a very widespread, accessible and easy-to-use telecommunication medium, to break down the geographical, logistical, socio-demographic and organizational barriers that make it difficult and/or prevent 1) access to these clinical services and 2) the continuity of their provision, as well as the creation and completion of 3) large-scale epidemiological studies and 4) decentralized clinical trials. However, although some TBCS tests have recently been developed and standardized in Italy, their clinimetric properties and clinical usability in populations with chronic neurological disorders have not yet been investigated. Furthermore, currently, the "paper-and-pencil" version of the international gold-standard for TBCS procedures . i.e. the Telephone Interview For Cognitive Status (TICS), which has been recently standardized in this country - is not available within the Italian scenario. In fact, although the feasibility of a de visu version of the TICS (i.e., In-Person TICS; IP-TICS) has been demonstrated in this country, an actual standardization of this test has not yet been implemented to date. Such a tool would, however, allow flexible use of screening assessments, regardless of the delivery method, both in clinical and experimental contexts.
2. Aims

   The present study primarily aims to provide exhaustive evidence regarding the psychometric, diagnostic and both cross-sectional and longitudinal clinical usability of TBCS that are currently available within the Italian scenario in populations with chronic neurological disorders. Secondly, this study aims to derive, in normotypical Italian subjects, 1) normative data for the IP-TICS and 2) the conversion algorithms between the latter (and other widely used "paper-and-pencil" screeners ) and the TICS.
3. Methods

The study is monocentric, observational, prospective. Over a period of 3 years, patients who have already undergone an in-person cognitive screening session within 6 months prior to recruitment and falling under the following diagnostic categories will be recruited: 1) amyotrophic lateral sclerosis (N≥88); 2) Alzheimer's disease (N≥66); 3) Lewy body dementia (N≥30); 4) frontotemporal dementia (N≥30); 5) chronic cerebrovascular disorders (N≥66). Furthermore, N≥287 normotypical subjects representative of the Italian population will be recruited. The following TBCS tests will be administered to patients: 1) TICS; 2) Telephone-based Frontal Assessment Battery; 3) Telephone Language Screener; 4) Telephone-based Verbal Fluency Battery; 5) ALS Cognitive Behavioral Screen-Phone Version. Additionally, patients will undergo a functional evaluation using caregiver-report questionnaires evaluating instrumental and non-instrumental skills of daily living and behavioral changes. Normal subjects will instead be administered: 1) TICS; 2) IP-TICS; 3) Mini-Mental State Examination (MMSE); 4) Montreal Cognitive Assessment (MoCA). In patients, telephone follow-ups are expected after 6, 12 and 18 months. Statistical analyses will be carried out aimed at 1) the detailed study, in patients, of the psychometrics, diagnostics and cross-sectional/longitudinal clinical usability of the aforementioned TBCS test, as well as at 2) the derivation, in normotypical subjects, of the normative data of the IP-TICS and MoCA Memory Index Score (MIS), as well as the conversion algorithms between TICS and IP-TICS/MMSE/MoCA.

ELIGIBILITY:
Inclusion criteria:

Patient cohorts: diagnosis of interest. NIs: not applicable

Exclusion Criteria:

Patient cohorts

* age <18 years;
* denial of informed consent to voluntary participation and data processing;
* absence of the diagnosis of interest;
* absence of a de visu cognitive screening assessment carried out in the 6 months prior to recruitment;
* positive history of 1) psychiatric pathologies, 2) serious and/or uncompensated general-medical conditions and 3) uncorrected visual/hearing deficits.

NIs:

* age <18 years;
* denial of informed consent to voluntary participation and data processing;
* positive history of 1) brain disorders, 2) serious and/or uncompensated general-medical conditions and 3) uncorrected visual/hearing deficits.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS: individuals having received a clinical diagnosis of ALS according to current diagnostic criteria AD: individuals with mild cognitive impairment/dementia due to either clinically- or neurochemically-confirmed Alzheimer's disease according to current diagnostic criteria LBD: individuals having received a clinical diagnosis of LBD according to current diagnostic criteria FTD: individuals having received a clinical diagnosis of FTD according to current diagnostic criteria CVD: individuals with mild cognitive impairment/dementia due to neuroradiologically-confirmed chronic cerebrovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
ALS Cognitive Behavioral Screen-Phone Version in ALS patients | At enrollment and at 6 months, 12 months and 18 months of follow-up
  ALS Cognitive Behavioral Screen-Phone Version
Telephone Interview for Cognitive Status in AD, LBD, FTD and CVD patients | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Telephone Interview for Cognitive Status
Telephone-based Frontal Assessment Battery in ALS, AD, LBD, FTD and CVD patients | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Telephone-based Frontal Assessment Battery
Telephone Language Screener in ALS, AD, LBD, FTD and CVD patients | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Telephone Language Screener
Telephone-based Verbal Fluency Battery in ALS, AD, LBD, FTD and CVD patients | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Telephone-based Verbal Fluency Battery
Mini-Mental State Examination in NI | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Mini-Mental State Examination; test with minimum score of 0 and maximum score of 30
Montreal Cognitive Assessment in NI | At enrollment and at 6 months, 12 months and 18 months of follow-up
  Montreal Cognitive Assessment; test with maximum score of 30: score of 26 or more is considered normal

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy